CLINICAL TRIAL: NCT06406894
Title: Effect of Superficial Back Line Relaxation Technique on Hamstring Flexibility in Non Specific Low Back Pain Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/MS-PT/01797
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Low Back Pain, Mechanical; Hamstring Flexibility
Keywords: hamstring flexibility; backache; Suboccipital muscle inhibition technique; cranial cervical flexion exercise
MeSH Terms: conditions — Low Back Pain; Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- superficial back line relaxation (Experimental): suboccipital muscle inhibition, cranial cervical flexion exercise
  Interventions: Other: Superficial back line relaxation (SMIT & CCFE)
- Conventional physical therapy (Active Comparator): hot packs, muscle stretching exercise of lowerlimb ( Pelvic bridging, knee to chest, Cat and camel stretch)
  Interventions: Other: Conventional physical therapy

INTERVENTIONS:
Other: Conventional physical therapy — lower limb muscle stretching ( pelvic bridging, Knee to chest,cat and camel stretch) (30 seconds hold and 3 sets of 5 repetitions with 1 min rest interval in between each set, per session on daily basis for only one week for immediate results and for long term effect on alternate 3 days in remaining 2nd ,3rd week).
  Treatment protocol will be given on daily basis to check immediate effect and for long term effect treatment will be given in alternating 3 days for remaining 2 weeks. Total 12 session were given (3 weeks).
  Arms: Conventional physical therapy
Other: Superficial back line relaxation (SMIT & CCFE) — Experimental group was given superficial back line relaxation includes SMIT & CCFE along with conventional therapy includes lower limb muscle stretching. SMIT For short term effect 10-12 repetitions per session, on daily basis for 1st week. For long term effect 10-12 repetitions per session, for 3 alternate days in remaining 2nd&3rd week. CCFE For short term effect 3 sets of 10 reps , 10 sec hold , 1 min rest after each set, on daily basis for 1st week. For long term effect 3 sets of 10 reps, 10 sec hold , 1 min rest after each set, for 3 alternate days , remaining 2nd & 3rd week. Conventional therapy lower limb muscle stretching ( For short term effect 30 seconds hold , 3 sets of 5 repetitions , 1 min rest after each set, per session on daily basis for 1st week , for long term effect on alternate 3 days in remaining 2nd ,3rd week). Total 12 sessions were given (3 weeks).
  Arms: superficial back line relaxation

SUMMARY:
Current study aim to evaluate the effect of Superficial back line relaxation techniques (SMIT along with CCFE) In Non Specific Low back Pain Patients in order to improve pain and hamstring flexibility.

And To find out the association between sub occipital muscle inhibition technique (SMIT) and cranial cervical flexion exercise (CCFE) in nonspecific low back pain patients with hamstring tightness.

The study aims to enhance the functional status and posture of patients suffering from nonspecific low back pain due to hamstring tightness, thereby enhancing patient efficiency in performing ADLS and IADLS.

DETAILED DESCRIPTION:
According to recent studies, hamstring tightness gets better as a result of sub occipital muscle inhibition technique, and cranial cervical flexion exercise that improve hamstring flexibility. SMIT is an approach of releasing fascia by application of pressure on sub occipital area. The myofascia relaxes as tone of suboccipital muscle declines that results in reduction in hamstring tone effectively.This is so because the superficial back line of dura matter connects hamstring with sub occipital muscles and neurological system runs through it. In SMIT superficial back line relaxes. While this approach helps suboccipital muscles release degree tension between occiput and axis.

The premise behind CCFE is that cervical spine's dura matter and suboccipital muscle fascia are connected by soft tissue while superficial back line of myofascial chain connects the neck to lower extremity. If tone of suboccipital muscle is reduced,the tone of knee flexors gets minimize and degree of hip flexion gets increase that results in increasing hamstring flexibility. Previous study showed that CCFE restores hamstring flexibility by relaxing superficial back line. While SMI and CCFE represents passive and active exercise program, respectively are equally effective in immediate enhancement of hamstring flexibility.

This study divide in to two groups. Group A ( experimental group) and Group B ( control group). Group A will receive manual technique superficial back line relaxation technique includes (Suboccpital muscle inhibition along with cranial cervical flexion Exercise) with conventional therapy.While group B will receive only conventional therapy include hot pack (lumber region) with low back exercises such as stretching exercise (knee to chest, Pelvis bridging, Cat and camel stretch).

Current study aims to pin point combine effect of SMIT along with CCFE in people with hamstring tightness. Additionally this study will evaluate the immediate and long term effect of SMIT and CCFE on patients with non- specific low back pain by comparing direct and indirect approaches for hamstring flexibility. The study aims to enhance the functional status and posture of patients suffering from nonspecific low back pain due to hamstring tightness, thereby enhancing patient efficiency in performing ADLS and IADLS.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic low back pain associate with hamstring tightness.
* Unilateral or bilateral short hamstring syndrome
* 3 to 6 points in numeric pain rating scale(NPRS).
* Active knee extension more than 20°.
* Presence of hamstring tightness with Popliteal angle more than 30 degree.
* Angle in SLR test should be less than 80°

Exclusion Criteria:

* History of cervical spine surgery and neck trauma.
* Cervical and lumber spinal deformity, Herniated disc or protrusions, Spinal stenosis.
* Muscle tendon injuries of the hamstring.
* History of vascular disease in head and neck.
* Visual swelling in the region of hamstring muscle.
* Progressive neurological deficit.
* Fractures in cervical and lumber spine.
* Past and current history of vertigo and dizziness.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Politeal angle ( Hip flexion with knee extension range) | 3rd week
  Changes from baseline popliteal angle was taken with help of goniometer. The hamstring-popliteal angle measures hamstring flexibility by bending the hip and stretching the knee. It's passive and accurate, with a 98% reliability value. Adult popliteal angles typically fall between 80 and 90 degrees. If leg cannot reach this angle, stiffness may be present.
Straight leg raise SLR (Hip flexion ROM) | 3rd week
  Changes from baseline hip flexion ROM was taken with help of goniometer. Patient lies supine throughout the SLR test, and the assessor raises the subject's right leg. Patient should keep their leg straight during the evaluation. If the therapist senses resistance or the patient complains of pain, the therapist should halt and use goniometry to determine the angle of the lower leg and hip. The therapist need to be vigilance while measuring the angle to make sure the patient's ankle or pelvis does not rotate. This test's reliability for determining hamstring flexibility is 92%.
Active knee extension test | 3rd week
  Changes from baseline knee extension range was taken with help of goniometer. This test was performed to assess the hamstring muscle's flexibility.The length of the hamstring muscles was determined by measuring the angle of knee extension in degrees. This test has a 99% reliability rate when used to measure hamstring flexibility
Modified Sit and Reach test | 3rd week
  Common test of flexibility that evaluates the hamstring and lower back muscles' flexibility is the sit and reach test.The greatest distance a person can extend forward while seated in a fixed position is measured, and this is used to evaluate the stability of the patient.The sit-and-reach test's reliability rate for hamstring flexibility is 96%.

SECONDARY OUTCOMES:
Numeric pain rating scale(NPRS) | 3rd week
  Changes from baseline NPRS is a one-dimensional assessment of adult pain severity, where participants rate their discomfort using a segmented numeric version (0-10 integers) of the VAS. NPRS has a 96% reliability rate and an 85% validity rate..
Oswestry Disability Index (ODI) | 3rd week
  (ODI) is a widely used tool for measuring low back pain, assessing impairment in daily activities. It uses a questionnaire with 10 multiple-choice questions.Each question contains six possible answers, ranging from 0 to 5, indicating a person's ability to perform specific tasks. ODI has a 96% reliability rate.

CONTACTS AND LOCATIONS:
Overall Officials: Sidra Ghais, Phd, Principal Investigator — Riphah International University
Locations (1):
- Railway General hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cho SH, Kim SH, Park DJ. The comparison of the immediate effects of application of the suboccipital muscle inhibition and self-myofascial release techniques in the suboccipital region on short hamstring. J Phys Ther Sci. 2015 Jan;27(1):195-7. doi: 10.1589/jpts.27.195. Epub 2015 Jan 9. PMID 25642072
- [Background] Houston MN, Hodson VE, Adams KK, Hoch JM. The effectiveness of whole-body-vibration training in improving hamstring flexibility in physically active adults. J Sport Rehabil. 2015 Feb;24(1):77-82. doi: 10.1123/JSR.2013-0059. PMID 25606860
- [Background] Strand SL, Hjelm J, Shoepe TC, Fajardo MA. Norms for an isometric muscle endurance test. J Hum Kinet. 2014 Apr 9;40:93-102. doi: 10.2478/hukin-2014-0011. eCollection 2014 Mar 27. PMID 25031677
- [Background] Coenen P, Gouttebarge V, van der Burght AS, van Dieen JH, Frings-Dresen MH, van der Beek AJ, Burdorf A. The effect of lifting during work on low back pain: a health impact assessment based on a meta-analysis. Occup Environ Med. 2014 Dec;71(12):871-7. doi: 10.1136/oemed-2014-102346. Epub 2014 Aug 27. PMID 25165395
- [Background] Simmonds N, Miller P, Gemmell H. A theoretical framework for the role of fascia in manual therapy. J Bodyw Mov Ther. 2012 Jan;16(1):83-93. doi: 10.1016/j.jbmt.2010.08.001. Epub 2010 Sep 27. PMID 22196432
- [Background] Massoud Arab A, Reza Nourbakhsh M, Mohammadifar A. The relationship between hamstring length and gluteal muscle strength in individuals with sacroiliac joint dysfunction. J Man Manip Ther. 2011 Feb;19(1):5-10. doi: 10.1179/106698110X12804993426848. PMID 22294848
- [Background] Jull GA, Falla D, Vicenzino B, Hodges PW. The effect of therapeutic exercise on activation of the deep cervical flexor muscles in people with chronic neck pain. Man Ther. 2009 Dec;14(6):696-701. doi: 10.1016/j.math.2009.05.004. Epub 2009 Jul 25. PMID 19632880
- [Background] Jeong ED, Kim CY, Kim SM, Lee SJ, Kim HD. Short-term effects of the suboccipital muscle inhibition technique and cranio-cervical flexion exercise on hamstring flexibility, cranio-vertebral angle, and range of motion of the cervical spine in subjects with neck pain: A randomized controlled trial. J Back Musculoskelet Rehabil. 2018;31(6):1025-1034. doi: 10.3233/BMR-171016. PMID 30248030
- [Background] Rogan S, Wust D, Schwitter T, Schmidtbleicher D. Static stretching of the hamstring muscle for injury prevention in football codes: a systematic review. Asian J Sports Med. 2013 Mar;4(1):1-9. Epub 2012 Nov 20. PMID 23785569
- [Background] Ajimsha MS, Daniel B, Chithra S. Effectiveness of myofascial release in the management of chronic low back pain in nursing professionals. J Bodyw Mov Ther. 2014 Apr;18(2):273-81. doi: 10.1016/j.jbmt.2013.05.007. Epub 2013 Jun 5. PMID 24725797
- [Background] Hart DL, Stratford PW, Werneke MW, Deutscher D, Wang YC. Lumbar computerized adaptive test and Modified Oswestry Low Back Pain Disability Questionnaire: relative validity and important change. J Orthop Sports Phys Ther. 2012 Jun;42(6):541-51. doi: 10.2519/jospt.2012.3942. Epub 2012 Apr 19. PMID 22517215